CLINICAL TRIAL: NCT02976987
Title: A Prolongation of Phase II Clinical Study to Evaluate the Efficacy of an Aqueous Gel Containing 2% (w/w) of Cidofovir, Directly Applied on the Cervix Exhibiting High Grade Squamous Intraepithelial Lesions
Brief Title: A Prolongation of a Clinical Study to Evaluate the Efficacy of an Aqueous Gel Containing 2% (w/w) of Cidofovir, Directly Applied on the Cervix Exhibiting High Grade Squamous Intraepithelial Lesions.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Catherine Vanpachterbeke, Head of clinic, Brugmann University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-POST-Colvir II
Record Dates: First submitted 2016-11-15; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: High Grade Cervical Epithelial Neoplasia (CIN2+)
Keywords: Colvir; high grade squamous intraepithelial lesions; cervix
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir (Experimental): Women receiving an aqueous gel containing 2% (w/w) cidofovir, administrated directly on cervix exhibiting high grade squamous intraepithelial lesion (CIN 2 and 3).
  Interventions: Drug: Cidofovir

INTERVENTIONS:
Drug: Cidofovir

SUMMARY:
The infections of high grade induced by the human papilloma viruses cause precancerous lesions of the cervical epithelium. The progression of these lesions can lead to the onset of cervical cancer. To reduce the risk of cancer lesions classified as 'cervical squamous intraepithelial neoplasia 2' (CIN2) and 'cervical squamous intraepithelial neoplasia 3' (CIN3), the standard treatment is the conisation of the cervix. This surgery can lead to complications such as infertility or a risk of preterm birth, hence the need to move towards a non-surgical alternative therapy.

The colvir clinical trial was a phase-II, multi center, randomized, double blind, efficacy study of an aqueous gel containing 2% (w/w) cidofovir, administrated directly on cervix exhibiting high grade squamous intraepithelial lesion (CIN 2 and 3).

This clinical trial is a prolongation of the colvir trial, in order to

* assess the long term histological and virological evolution (24 months) of 3 g of 2% (w/w) cidofovir gel, administrated directly on cervix exhibiting high grade intraepithelial neoplasia after complete response, partial response or response failure at the end of the Colvir study.
* assess the long term (24 months) rate of recurrence of histological lesions of the Colvir patients after conisation, in both placebo and treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Women who participated in the COLVIR study and received complete treatment

Exclusion Criteria:

* Women from the Colvir study who received incomplete treatment

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
change in biopsy conclusions (treatment success or not) | 24 months after initial treatment
  A gynecological examination will be done, including colposcopy. Cervical sampling for virology will be taken and sent to Riatol laboratory. A biopsy will be taken in presence of colposcopic cervical squamous intraepithelial neoplasia (CIN2-3) lesions, or in case of colposcopic doubt lesions, or in case of persistence (after 6 months) of colposcopic CIN1 lesion or if the last cytology was a high grade squamous intraepithelial lesion (HSIL) cytology, or if the last cytology suspected glandular lesions, or if the two last cervical smears were low-grade intraepithelial lesion (LSIL) cytologies with presence of high risk human papillomavirus (HPV).The biopsy fixation, HE (eosin-hematoxylin) staining and P16 + Ki67 staining will be done according to a validated procedure. Biopsy slides will be send to the central lab for immunological and histological reading (three pathologic experts).

SECONDARY OUTCOMES:
HPV viral load | 24 months after initial treatment
  Cervical sampling for virology will be taken and send to Riatol laboratory.
HPV genotype | 24 months after initial treatment
  Cervical sampling for virology will be taken and send to Riatol laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Vanpachterbeke, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann Hospital, Brussels, Belgium